CLINICAL TRIAL: NCT03519854
Title: A Multi-center, Randomized, Assessor-blinded, Placebo Controlled, Phase II, Parallel Dose-finding Trial in Male Subjects of ASA 1-2 to Assess the Efficacy, Safety and Pharmacokinetics of 5 Doses of Org 25969 When Administered After 0.6 mg.Kg-1 Esmeron® at 3, 5 or 15 Minutes
Brief Title: Efficacy, Safety and Pharmacokinetics of Sugammadex (Org 25969; MK-8616) at 3 Different Time Points After 0.6 mg/kg Esmeron® in Male Participants (P05940; MK-8616-020).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P05940; MK-8616-020 (Other: Merck Protocol Number); 19.4.202 (Other: Organon Protocol Number)
Record Dates: First submitted 2018-05-08; First posted 2018-05-09 (Actual); Results first posted 2019-02-01 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (18):
- Arm A. Placebo; given 3 minutes after Esmeron® (Placebo Comparator): Placebo (single intravenous (IV) bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm B. 1 mg/kg Sugammadex; given 3 minutes after Esmeron® (Experimental): Sugammadex (1 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm C. 2 mg/kg Sugammadex; given 3 minutes after Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm D. 4 mg/kg Sugammadex; given 3 minutes after Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm E. 6 mg/kg Sugammadex; given 3 minutes after Esmeron® (Experimental): Sugammadex (6 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm F. 8 mg/kg Sugammadex; given 3 minutes after Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm G. Placebo; given 5 minutes after Esmeron® (Placebo Comparator): Placebo (single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm H. 1 mg/kg Sugammadex; given 5 minutes after Esmeron® (Experimental): Sugammadex (1 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm I. 2 mg/kg Sugammadex; given 5 minutes after Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm J. 4 mg/kg Sugammadex; given 5 minutes after Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm K. 6 mg/kg Sugammadex; given 5 minutes after Esmeron® (Experimental): Sugammadex (6 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm L. 8 mg/kg Sugammadex; given 5 minutes after Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm M. Placebo; given 15 minutes after Esmeron® (Placebo Comparator): Placebo (single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Placebo; Drug: Esmeron®
- Arm N. 1 mg/kg Sugammadex; given 15 minutes after Esmeron® (Experimental): Sugammadex (1 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm O. 2 mg/kg Sugammadex; given 15 minutes after Esmeron® (Experimental): Sugammadex (2 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm P. 4 mg/kg Sugammadex; given 15 minutes after Esmeron® (Experimental): Sugammadex (4 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm Q. 6 mg/kg Sugammadex; given 15 minutes after Esmeron® (Experimental): Sugammadex (6 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®
- Arm R. 8 mg/kg Sugammadex; given 15 minutes after Esmeron® (Experimental): Sugammadex (8 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
  Interventions: Drug: Sugammadex; Drug: Esmeron®

INTERVENTIONS:
Drug: Placebo — 0.9% NaCl administered as a fast IV bolus dose (within 30 seconds).
  Arms: Arm A. Placebo; given 3 minutes after Esmeron®; Arm G. Placebo; given 5 minutes after Esmeron®; Arm M. Placebo; given 15 minutes after Esmeron®
Drug: Sugammadex — Sugammadex administered as a fast IV bolus dose (within 30 seconds), dosed according to participant actual body weight.
  Other Names: Org 25969; MK-8616; Bridion®.
  Arms: Arm B. 1 mg/kg Sugammadex; given 3 minutes after Esmeron®; Arm C. 2 mg/kg Sugammadex; given 3 minutes after Esmeron®; Arm D. 4 mg/kg Sugammadex; given 3 minutes after Esmeron®; Arm E. 6 mg/kg Sugammadex; given 3 minutes after Esmeron®; Arm F. 8 mg/kg Sugammadex; given 3 minutes after Esmeron®; Arm H. 1 mg/kg Sugammadex; given 5 minutes after Esmeron®; Arm I. 2 mg/kg Sugammadex; given 5 minutes after Esmeron®; Arm J. 4 mg/kg Sugammadex; given 5 minutes after Esmeron®; Arm K. 6 mg/kg Sugammadex; given 5 minutes after Esmeron®; Arm L. 8 mg/kg Sugammadex; given 5 minutes after Esmeron®; Arm N. 1 mg/kg Sugammadex; given 15 minutes after Esmeron®; Arm O. 2 mg/kg Sugammadex; given 15 minutes after Esmeron®; Arm P. 4 mg/kg Sugammadex; given 15 minutes after Esmeron®; Arm Q. 6 mg/kg Sugammadex; given 15 minutes after Esmeron®; Arm R. 8 mg/kg Sugammadex; given 15 minutes after Esmeron®
Drug: Esmeron® — Esmeron® administered at 0.6 mg/kg as a fast IV bolus (within 10 seconds), dosed according to participant actual body weight.
  Other Names: Rocuronium bromide

SUMMARY:
This study investigates the efficacy, safety, and pharmacokinetics of sugammadex (Org 25969; MK-8616) when administered for the reversal of neuromuscular blockade in male participants receiving surgery, classified as American Society of Anesthesiologists (ASA) class 1 (otherwise normal, healthy participant) to class 2 (participant with mild systemic disease). The primary objective of this study is to explore the dose-response relation of sugammadex given as a reversal agent at 3, 5, or 15 minutes following administration of 0.6 mg/kg Esmeron®.

ELIGIBILITY:
Inclusion Criteria:

* Participants of ASA class 1 to 2.
* Participants scheduled for surgical procedures with an anticipated duration of anesthesia of at least 75 minutes, without further need for muscle relaxation other than for intubation.

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations is expected.
* Participants known or suspected to have neuromuscular disorders and/or significant hepatic or renal dysfunction.
* Participants known or suspected to have a (family) history of malignant hyperthermia.
* Participants known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia.
* Participants receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants, aminoglycosides, and Mg^2+.
* Participants who have already participated in this trial.
* Participants who have participated in another clinical trial, not pre-approved by NV Organon, within 30 days of entering into this trial.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2002-12-01 (Actual); Primary Completion 2003-06-01 (Actual); Study Completion 2003-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the N=99 randomized participants, N=98 received treatment. Treated participants are counted as Started in the arm that most accurately describes the treatment received. If no treatment was received (N=1 participant), participants are counted as Started in the arm to which they were randomized.
Pre-assignment Details: One participant originally randomized to receive 2 mg/kg Sugammadex, given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. As a result, this participant is counted as Started/Treated in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Period: Overall Study
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Started | 4 (N=3 randomized to Arm A. An additional N=1 (randomized to Arm C) is counted as Started in Arm A) | 6 | 5 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
Treated | 4 (N=1 (randomized to Arm C) received placebo, 3 min after 1.2 mg/kg Esmeron®) | 6 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
Completed | 4 | 6 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Technical Error | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all randomized participants receiving study treatment. One participant randomized to receive 2 mg/kg Sugammadex, given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Total
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Includes all randomized participants receiving study treatment. One participant randomized to receive 2 mg/kg Sugammadex, given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
  Years | 49.8 (12.1) | 35.5 (14.0) | 35.8 (16.2) | 41.3 (11.6) | 34.3 (9.3) | 39.0 (7.7) | 38.7 (18.6) | 35.0 (11.5) | 40.5 (12.4) | 40.8 (8.4) | 38.7 (11.9) | 31.5 (11.8) | 33.0 (5.6) | 48.3 (11.6) | 39.8 (17.2) | 41.7 (13.6) | 36.0 (12.1) | 40.2 (15.8) | 38.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Includes all randomized participants receiving study treatment. One participant randomized to receive 2 mg/kg Sugammadex, given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Male | 4 | 6 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mean Time From Start of Study Treatment Administration to Recovery of the T4/T1 Ratio to 0.9
Description: Mean time from start of study treatment administration to recovery of participant T4/T1 ratio to 0.9 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of neuromuscular blockade (NMB) present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.9 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to 70 minutes following administration of study treatment
Population: Per protocol, includes all randomized participants receiving study treatment without major protocol violations, having data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 5 | 5 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
minutes | 52.05 (8.77) | 22.73 (11.58) | 4.93 (1.25) | 6.25 (9.00) | 1.85 (0.62) | 1.83 (0.87) | 51.67 (13.13) | 27.35 (6.35) | 8.88 (7.80) | 2.28 (0.73) | 2.13 (0.93) | 1.45 (0.60) | 35.58 (9.05) | 6.53 (1.73) | 2.73 (0.72) | 2.05 (1.18) | 2.08 (1.97) | 1.35 (0.20)

2. Secondary Outcome: Mean Heart Rate at Baseline
Description: Mean heart rate at baseline was assessed. Baseline heart rate was defined as the heart rate measured under stable anesthesia prior to administration of study treatment.
Time Frame: Up to 45 minutes prior to study treatment administration
Population: All randomized participants receiving study treatment, having data available at baseline prior to administration of study treatment. One participant randomized to receive 2 mg/kg Sugammadex, given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
beats per minute (bpm) | 61.0 (3.6) | 62.0 (4.6) | 63.5 (3.9) | 68.0 (11.4) | 68.2 (10.8) | 69.8 (18.5) | 68.0 (10.6) | 56.7 (10.9) | 64.2 (10.5) | 64.7 (7.2) | 69.7 (21.0) | 57.5 (4.7) | 63.0 (11.8) | 62.7 (8.8) | 65.3 (13.5) | 64.2 (8.6) | 66.5 (11.7) | 68.5 (9.4)

3. Secondary Outcome: Mean Heart Rate at 2 Minutes Following Administration of Study Treatment
Description: Mean heart rate at 2 minutes following administration of study treatment was assessed.
Time Frame: 2 minutes following administration of study treatment
Population: All randomized participants receiving study treatment, having data available at 2 minutes following administration of study treatment. One participant randomized to receive 2 mg/kg Sugammadex at 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 5 | 6 | 3 | 6 | 6 | 6 | 5 | 6 | 2 | 5 | 5 | 6 | 5 | 6
bpm | 76.7 (18.6) | 73.0 (15.0) | 84.5 (12.0) | 72.7 (12.1) | 86.2 (15.5) | 74.8 (17.7) | 84.0 (15.1) | 61.3 (11.2) | 70.8 (13.7) | 66.2 (9.8) | 69.8 (21.3) | 67.8 (10.2) | 59.0 (1.4) | 71.2 (12.9) | 77.2 (16.5) | 62.8 (5.0) | 65.4 (14.7) | 64.3 (5.4)

4. Secondary Outcome: Mean Heart Rate at 30 Minutes Following Administration of Study Treatment
Description: Mean heart rate at 30 minutes following administration of study treatment was assessed.
Time Frame: 30 minutes following administration of study treatment
Population: All randomized participants receiving study treatment, having data available at 30 minutes following administration of study treatment. One participant randomized to receive 2 mg/kg Sugammadex at 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 6 | 5 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
bpm | 77.8 (8.6) | 62.0 (2.8) | 72.0 (7.8) | 72.5 (9.6) | 76.7 (11.2) | 66.6 (15.2) | 77.3 (9.5) | 63.0 (12.6) | 69.7 (11.4) | 72.5 (17.1) | 66.5 (23.9) | 60.0 (4.0) | 65.7 (16.8) | 66.8 (11.5) | 65.3 (10.8) | 63.5 (7.9) | 64.7 (14.3) | 66.0 (5.8)

5. Secondary Outcome: Mean Corrected QT Interval (QTc) at Baseline
Description: Mean QTc interval at baseline was assessed. Baseline QTc interval was defined as the QTc interval measured under stable anesthesia prior to administration of study treatment. The baseline QTc interval is corrected for participant heart rate at baseline prior to study treatment administration using Fridericia's correction, where QTc = QT interval/(RR interval)^(1/3). RR interval = 60/heart rate.
Time Frame: Up to 45 minutes prior to study treatment administration
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
milliseconds (msec) | 418 (2.5) | 396 (11.3) | 418 (17.8) | 404 (20.7) | 417 (13.1) | 416 (20.4) | 400 (23.9) | 415 (19.6) | 405 (15.7) | 416 (21.7) | 408 (22.2) | 411 (13.9) | 392 (13.9) | 410 (11.8) | 398 (14.5) | 398 (23.6) | 398 (24.8) | 406 (25.4)

6. Secondary Outcome: Mean Corrected QT Interval (QTc) at 2 Minutes Following Administration of Study Treatment
Description: Mean QTc interval at 2 minutes following administration of study treatment was assessed. The QTc interval is corrected for participant heart rate at 2 minutes following study treatment administration using Fridericia's correction, where QTc = QT interval/(RR interval)^(1/3). RR interval = 60/heart rate.
Time Frame: 2 minutes following administration of study treatment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 3 | 5 | 4 | 6 | 5 | 6 | 3 | 6 | 6 | 6 | 5 | 6 | 2 | 5 | 5 | 6 | 5 | 6
msec | 420 (13.7) | 406 (11.8) | 422 (17.0) | 406 (24.7) | 427 (10.5) | 416 (14.5) | 400 (27.5) | 420 (16.3) | 412 (16.6) | 419 (20.3) | 410 (24.9) | 416 (20.2) | 401 (4.2) | 419 (15.6) | 406 (12.9) | 416 (26.5) | 410 (31.8) | 416 (16.8)

7. Secondary Outcome: Mean Corrected QT Interval (QTc) at 30 Minutes Following Administration of Study Treatment
Description: Mean QTc interval at 30 minutes following administration of study treatment was assessed. The QTc interval is corrected for participant heart rate at 30 minutes following study treatment administration using Fridericia's correction, where QTc = QT interval/(RR interval)^(1/3). RR interval = 60/heart rate.
Time Frame: 30 minutes following administration of study treatment
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 4 | 4 | 4 | 6 | 6 | 5 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
msec | 418 (11.6) | 416 (17.6) | 427 (13.2) | 415 (21.7) | 433 (21.6) | 424 (27.0) | 392 (21.1) | 420 (21.3) | 425 (19.6) | 413 (21.9) | 400 (27.4) | 422 (14.4) | 400 (6.8) | 418 (18.5) | 408 (14.6) | 421 (33.8) | 411 (25.3) | 418 (22.0)

8. Secondary Outcome: Number of Participants Experiencing an Adverse Event
Description: The number of participants experiencing an adverse event (AE) was assessed. An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product.
Time Frame: Up to 7 days following administration of study treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron® | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron® | Arm G. Placebo; Given 5 Minutes After Esmeron® | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron® | Arm M. Placebo; Given 15 Minutes After Esmeron® | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron® | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron®
Number analyzed (Participants) | 4 | 6 | 4 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 5 | 1 | 4 | 4 | 5 | 2 | 2 | 1 | 3 | 2 | 2 | 0 | 4 | 4 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 7 days following administration of study treatment
Description: Includes all randomized participants receiving study treatment. One participant randomized to receive 2 mg/kg Sugammadex given 3 minutes after Esmeron® (Arm C), incorrectly received placebo. This participant is counted in the "Arm A. Placebo; given 3 minutes after Esmeron®" arm.
Groups:
- Arm A. Placebo; Given 3 Minutes After Esmeron: Placebo (single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron: Sugammadex (1 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron: Sugammadex (6 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 3 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm G. Placebo; Given 5 Minutes After Esmeron: Placebo (single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron: Sugammadex (1 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron: Sugammadex (6 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 5 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm M. Placebo; Given 15 Minutes After Esmeron: Placebo (single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron: Sugammadex (1 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron: Sugammadex (2 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron: Sugammadex (4 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron: Sugammadex (6 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
- Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron: Sugammadex (8 mg/kg; single IV bolus) administered 15 minutes after the bolus intubation dose of 0.6 mg/kg Esmeron®.
Arm/Group | Arm A. Placebo; Given 3 Minutes After Esmeron | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron | Arm G. Placebo; Given 5 Minutes After Esmeron | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron | Arm M. Placebo; Given 15 Minutes After Esmeron | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/4 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 5/6 | 1/4 | 4/6 | 4/6 | 5/6 | 2/3 | 2/6 | 1/6 | 3/6 | 2/6 | 2/6 | 0/3 | 4/6 | 4/6 | 1/6 | 1/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A. Placebo; Given 3 Minutes After Esmeron (N=4) | Arm B. 1 mg/kg Sugammadex; Given 3 Minutes After Esmeron (N=6) | Arm C. 2 mg/kg Sugammadex; Given 3 Minutes After Esmeron (N=4) | Arm D. 4 mg/kg Sugammadex; Given 3 Minutes After Esmeron (N=6) | Arm E. 6 mg/kg Sugammadex; Given 3 Minutes After Esmeron (N=6) | Arm F. 8 mg/kg Sugammadex; Given 3 Minutes After Esmeron (N=6) | Arm G. Placebo; Given 5 Minutes After Esmeron (N=3) | Arm H. 1 mg/kg Sugammadex; Given 5 Minutes After Esmeron (N=6) | Arm I. 2 mg/kg Sugammadex; Given 5 Minutes After Esmeron (N=6) | Arm J. 4 mg/kg Sugammadex; Given 5 Minutes After Esmeron (N=6) | Arm K. 6 mg/kg Sugammadex; Given 5 Minutes After Esmeron (N=6) | Arm L. 8 mg/kg Sugammadex; Given 5 Minutes After Esmeron (N=6) | Arm M. Placebo; Given 15 Minutes After Esmeron (N=3) | Arm N. 1 mg/kg Sugammadex; Given 15 Minutes After Esmeron (N=6) | Arm O. 2 mg/kg Sugammadex; Given 15 Minutes After Esmeron (N=6) | Arm P. 4 mg/kg Sugammadex; Given 15 Minutes After Esmeron (N=6) | Arm Q. 6 mg/kg Sugammadex; Given 15 Minutes After Esmeron (N=6) | Arm R. 8 mg/kg Sugammadex; Given 15 Minutes After Esmeron (N=6)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Therapeutic response decreased (General disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (2) | 1 (3) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigators to publish, but all publications must be based on data validated by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.